CLINICAL TRIAL: NCT06240377
Title: Study of the Effectiveness of Percutaneous Neuromodulation and Transcranial Direct Current Stimulation vs Pharmacological Treatment in Cancer Patients With Lower Limb Pain
Brief Title: Effectiveness of NMP and TDCS vs Pharmacological Treatment in Cancer Patients With Lower Limb Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Canarias (Other)
Responsible Party: Principal Investigator, Eduardo Luis Martín Javier, Master of Science Professor Eduardo Martín, Universidad Europea de Canarias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22109-1
Record Dates: First submitted 2023-12-26; First posted 2024-02-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pain Cancer
Keywords: Cancer; Pain; Lower limb; TDCS; NMP
MeSH Terms: conditions — Cancer Pain; Neoplasms; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Simple Blind, Evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epte Bipolar System 2.0 - Ultrasound-guided percutaneous neuromodulation (NMP) (Active Comparator): EPTE Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system. Ultrasound-guided percutaneous neuromodulation (NMP)
  Interventions: Device: Ultrasound-guided percutaneous neuromodulation (NMP)
- Epte Bipolar System 2.0 - Transcranial direct current stimulation (tDCS) (Active Comparator): EPTE Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system. Transcranial direct current stimulation (tDCS)
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — EPTE Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system.
  It is a nationally manufactured device that meets all quality standards, being the perfect tool for the application of techniques such as tDCS. It is a versatile, compact, portable and easy to use equipment that has the ability to adapt the parameters to achieve any protocol established by scientific evidence to treat the various pathologies.
  The EPTE® Bipolar System device has an CE Health Certificate.
  Arms: Epte Bipolar System 2.0 - Transcranial direct current stimulation (tDCS)
Device: Ultrasound-guided percutaneous neuromodulation (NMP) — EPTE Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system.
  It is a nationally manufactured device that meets all quality standards, being the perfect tool for the application of techniques such as tDCS. It is a versatile, compact, portable and easy to use equipment that has the ability to adapt the parameters to achieve any protocol established by scientific evidence to treat the various pathologies.
  The EPTE® Bipolar System device has an CE Health Certificate.
  Arms: Epte Bipolar System 2.0 - Ultrasound-guided percutaneous neuromodulation (NMP)

SUMMARY:
the goal of this clinical trial is to compare in cancer patients:

Is ultrasound-guided percutaneous neuromodulation useful for lower limb pain relief in cancer patients?

Is direct current transcranial stimulation useful for relieving lower limb pain in cancer patients?

Participants will recive treatments of ultrasound-guided percutaneous neuromodulation and DC Transcranial Stimulation

Researchers will compare ultrasound-guided percutaneous neuromodulation and DC Transcranial Stimulation to see if pain in the lower extremities is reduced

DETAILED DESCRIPTION:
Increasing life expectancy, aging populations, and unhealthy lifestyles increase the likelihood of cancer. Lower limb pain is one of the most common symptoms causing functional incapacitation that makes it necessary to seek and improve its assessment tools, prevention and treatment.

Ultrasound-guided Percutaneous Neuromodulation is a technique that is being applied clinically by physical therapists. It is an accessible, minimally invasive, safe and economical procedure to apply.

Transcranial direct current stimulation is a non-invasive neuromodulation technique that has been widely studied for the treatment of chronic pain. It is an accessible, non-invasive, safe and cost-effective procedure to apply.

Traditional therapies have been, are and will continue to be useful tools to consider. The reduction in the manufacturing costs of assessment and treatment tools in recent years makes it affordable to obtain these equipment as intervention tools, since its usefulness in improving functionality and reducing pain is proven.

Opioid analgesics are the main tool for the treatment of pain in cancer patients, but adverse effects or inadequate treatment make necessary the search for other therapeutic tools more economical, rapid and with less risk of addiction and / or side effects.

Objective knowledge of the changes produced by this treatment and the ability to quantify the variation in pain suffered by patients becomes urgent to take steps forward in improving these symptoms.

Ultrasound evaluation has been confirmed as a useful tool to assess changes in tissue in a non-invasive, fast and safe way. Its high reliability has been widely proven.

Myotonometry has been consolidated in the last decade as a non-invasive assessment tool able to analyze the contractile properties of soft tissue quickly and safely. Its reliability has been validated in multiple studies.

For this reason, researchers propose to conduct research that improves and provides new data on its effectiveness and efficacy in the treatment of ultrasound-guided Percutaneous Neuromodulation and transcranial direct current stimulation therapy (tDCS).

ELIGIBILITY:
Inclusion Criteria:

The proposed inclusion criteria for the study are as follows:

* Age between 18 and 65.
* Pain in lower limbs
* Taking drug therapy for lower-extremity pain.
* Diagnosis of painful pathology in the anterior aspect of the knee secondary oncologic.

Exclusion Criteria:

The exclusion criteria are:

* Traumatic history
* Have had any type of analgesic treatment in the last 4 weeks (clinical, physical or orthostatic)
* No need for drug treatment within the last 30 days of study initiation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 12 weeks
  Numerical Pain Rating Scale (NPRS) Lower limb pain changes
  To mark its intensity patients should mark taking into account that 0 represents absence of pain and 10 the maximum pain imagined by the patient
Victorian Institute of Sport Assessment-Patella (VISA-P) | 12 weeks
  The VISA-P questionnaire is used for assessing the severity of symptoms in individuals with patellar tendinopathy, the term pain refers to the specific area of the patellar tendon, to mark its intensity patients should mark taking into account that 0 represents absence of pain and 10 the maximum pain imagined by the patient. In the analysis of patellar tendon pathology has already been used in repeated articles
OKS (Oxford Knee Score) | 12 weeks
  The Oxford Knee Score is a well-known tool for assessing quality of life in patients with Osteo Arthritis of the knee (OA). The OKS is a self-administered questionnaire that the patient can answer in face-to-face interviews or send by mail once completed. It contains 12 questions with 5 possible answers each aimed at evaluating the perception of the quality of life of the patient in the last four weeks. Each answer receives a score of 0 to 4, where 4 is the best possible result. After the sum, you get a total score ranging from 0 to 48, where 48 is the best possible result. The Spanish adaptation of the OKS questionnaire is a reliable tool to evaluate the perception of health-related quality of life of patients with knee osteoarthritis (KO)
Lower Limb functional Index (LLFFI) | 12 weeks
  The questionnaire contains a number of phrases (25 in total) that patients use to describe problems on their legs. Evaluating only the last few days if a phrase describes you should check that box, you can also mark it partially and if not you should leave it blank. Finally, an LLFI score is obtained where the functional index of the lower extremities is determined. The LLFI consists of 25 items with three-point response options (Yes = 1 point), ("In part" or "half" 1/2 points) and (NO Points = 0). With a gross score range of 0 to 25 points. Takes approximately 2 minutes. The score is calculated by simply adding the answers together and multiplying them by four minus 100 to convert them into a percentage scale or maximum loss of function. The LLFI questionnaire in Spanish proved to be suitable for assessing the functionality of the lower limbs and viable for the evaluation of the condition and deterioration of the lower limbs in clinical and research settings
RPE (Rating Perceived Exertion) | 12 weeks
  Borg created Borg's 15-point RPE scale. The modified RPE scale is 6 to 20 points. The level of physical exertion or perceived exertion is measured using the Borg 15-point RPE scale. A significant correlation was found between heart rate and Borg RPE of 15 points. In addition, this scale is thought to be a useful and economical tool for monitoring exercise intensity. Patients in clinical practice are instructed to choose a number from the scale and assess their total effort during endurance training. A score of six indicates lack of effort, or rest, and a score of twenty indicates maximum effort, or the most exhausting exercise
Threshold of pressure pain | 12 weeks
  The intensity of pain can provide relevant information, until now the measurement of pain was carried out subjectively for this reason there are efforts to develop devices to measure the intensity of painful stimuli objectively. Severity of pain also affects the patient's treatment strategy and goals because pain can cause incapacitation. Thus, several researchers have focused their efforts on creating pain-measuring devices called algometers. To measure this sensation, a pressure pain threshold (UDP)81 is usually used. It is applied at the above point and measured in N.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martín, Principal Investigator — Universidad Europea de Canarias
Locations (1):
- Centro RED Tenerife, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No